CLINICAL TRIAL: NCT04270903
Title: EPR (Electron Paramagnetic Resonance) as Method of Non-invasive Characterization of Melanin Content in Skins With Different Phototypes
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: MELA-RPE-PHOTOTYPE
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Skin Pigmentation; Free Radicals; Phototype; Magnetic Resonance
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phototype I - II: EPR measurement at the surface of the skin (arm)
  Interventions: Device: EPR measurement
- Phototype III - IV: EPR measurement at the surface of the skin (arm)
  Interventions: Device: EPR measurement
- Phototype V - VI: EPR measurement at the surface of the skin (arm)
  Interventions: Device: EPR measurement

INTERVENTIONS:
Device: EPR measurement — Subject put in a magnet, magnetic field sweeping around 40 mTesla. Irradiation with a wave with a frequency of 1.1 GHz. A resonator (surface coil) is put at the surface of the skin (arm). The EPR signal is recorded.

SUMMARY:
The aim of this study is to assess the signal of melanin using Electron Paramagnetic resonance (EPR). Melanin is a paramagnetic pigment detectable by EPR. Recent advances in instrumentation allows the application of EPR in human beings. The characterization of melanin by EPR could be potentially interesting in the context of melanoma detection and characterization. While another clinical study is currently ongoing aiming at demonstrating the feasibility of the non-invasive detection of the EPR signal of melanin in melanoma patients, it is crucial to have a control group with healthy skin. The aim of the present study is to assess the influence of skin pigmentation of the EPR signal recorded. In the present clinical study, the EPR signal of melanin will be characterized in healthy skin with different phototypes (1-2, 3-4, 5-6) to assess the potential influence of skin pigmentation on the EPR signal.

DETAILED DESCRIPTION:
Electron paramagnetic resonance (EPR), also known as electron spin resonance (ESR), is a spectrometric method enabling the observation of the absorption of energy by the free radicals contained by a sample immerged in a strong homogenous magnetic field. An EPR spectrum reveals only the presence of paramagnetic centers and can thus only be observed with samples containing lone unpaired electrons. In water-containing biological environments, most of free radicals are very reactive and have a very short life. To detect such species, a strategy is to use extrinsic molecules that will react with these species to form EPR measurable adducts. This technique is called "spin trapping". In contrast, the study of stable free radicals does not require the use of spin-trap agents. Melanins are part of the rare stable biological radicals directly observable with EPR. In practice, melanin is the only endogenous stable radical that can be detected using 1 GHz EPR.

The aim of the present study is to measure the EPR signal recorded from skin with different pigmentations. 45 healthy volunteers will be enrolled:

15 subjects with phototype 1-2, 15 subjects with phototypes 3-4, 15 subjects with phototypes 5-6. The parameters described hereafter will be investigated:

* g factor (resonance condition); expected g=2.005;
* shape of the signal, presence of a shoulder at g=2.01 due to pheomelanin;
* intensity of the signal (signal height, double integration, double integration relative to reference).

This will provide a database for other ongoing studies carried out in patients with suspicious lesion (nevi vs melanoma)

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with skin belonging to Phototype I-II, III-IV, V-VI

Exclusion Criteria:

* Subjects under 18 years
* Subjects with pacemakers
* Subjects with non-removable implants with metal or otherwise not known to be MRI-compatible.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 45 healthy volunteers
  * 15 subjects with skin Phototype I-II
  * 15 subjects with Phototype III-IV
  * 15 subjects with Phototype V-VI
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Measurement of the EPR signal intensity | Through study completion (6 months)
  Signal height / Double integration / Double integration relative to reference signal

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Gallez, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No